CLINICAL TRIAL: NCT00512070
Title: Melatonin Metabolism Abnormality in Patients With Schizophrenia or Schizoaffective Disorder Treated With Olanzapine and Melatonin Dose Finding for the Correction of the Metabolic Abnormality
Brief Title: Melatonin Metabolism Abnormality in Patients With Schizophrenia or Schizoaffective Disorder Treated With Olanzapine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F1D-MC-X302
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Results first posted 2024-12-05 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Obesity; Metabolic Syndrome
Keywords: schizophrenia; schizoaffective disorder; bipolar disorder; olanzapine; melatonin; obesity; metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Obesity; Metabolic Syndrome | interventions — Olanzapine; Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IIA (0.3mg day melatonin) (Experimental): 0.3mg day melatonin
  Interventions: Drug: olanzapine and melatonin
- IIB (3.0 mg/day melatonin) (Experimental): 3.0 mg/day melatonin
  Interventions: Drug: olanzapine and melatonin

INTERVENTIONS:
Drug: olanzapine and melatonin — In treatment phase I, all subjects will receive olanzapine, 10-25 mg/day. In treatment phase II, all subjects will receive olanzapine (10-25 mg/day) plus melatonin. Subjects will be randomized at a ratio of 1:1 to receive melatonin, 0.3 mg/day or 3.0 mg/day. Group IIA will receive 0.3mg day melatonin. Group IIB will receive 3.0 mg/day melatonin.
  Other Names: Olanzapine (Zyprexa)

SUMMARY:
Atypical antipsychotic medications, such as olanzapine, cause metabolic side effects, including weight gain, extra fat around the middle of the body, high blood sugar, and high cholesterol. One of the mechanisms by which these medications may cause these effects is by reducing plasma melatonin. This study is a pilot project to evaluate 1) the effect of olanzapine on melatonin secretion levels and 2) the effect of melatonin on olanzapine-induced changes in melatonin secretion in patients with schizophrenia, schizoaffective, or bipolar disorder.

DETAILED DESCRIPTION:
To investigate the relationship between olanzapine, melatonin, and metabolic functioning, this pilot study is evaluating 20 patients with schizophrenia, schizoaffective disorder, or bipolar disorder over 15 weeks under three experimental conditions: 1) baseline (two weeks treatment with already established antipsychotic medication other than olanzapine or clozapine), 2) six weeks treatment with olanzapine only, and 3) six weeks treatment with olanzapine and melatonin. Half of the patients will receive 0.3 mg of oral melatonin and half will receive 3.0 mg of melatonin. Nocturnal melatonin production, as estimated by assay of urinary 6-sulfatoxymelatonin(aMT6s) adjusted for creatinine, will be measured weekly. In addition, weekly measurements of weight and other metabolic indices, including waist and hip measurements, fasting glucose, serum insulin, cholesterol, triglycerides, and leptin will be taken. It is anticipated that there will be an olanzapine-induced decrease in melatonin production. Furthermore, it is expected that the decrease in melatonin production associated with olanzapine treatment will be reversed by administration of melatonin with olanzapine.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65;
2. DSM-IV-TR diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder;
3. Patients who, in the clinical judgment of the investigator, may benefit from a switch to olanzapine;
4. Females must be of non-child bearing potential (i.e., surgically sterilized, or at least one year post-menopausal) or on an appropriate dose of oral/depot contraceptives or using barrier protection and not breast-feeding. Females must have a urine pregnancy test at screening;
5. Willingness and ability to take medications nightly at 10:00 p.m.; and
6. The subject or his/her legal representative must provide informed, written consent.

Exclusion Criteria:

1. Females who are pregnant or lactating;
2. Concurrent participation or participation within the prior 30 days in any study involving investigational medications;
3. Current (within the prior 30 days) diagnosis of substance abuse or dependence;
4. Use of olanzapine within the prior three months;
5. History of allergy or intolerable side-effects to olanzapine in the past;
6. History of significant head trauma, defined as head trauma resulting in loss of consciousness for more than five minutes and/or neurological or cognitive sequelae;
7. Evidence of any clinically relevant disease (e.g., renal or hepatic impairment, significant coronary artery disease, cerebrovascular disease, or cancer) or any clinical finding that in the opinion of the investigator could potentially be negatively affected by study participation or that could potentially affect study participation is criterion for exclusion from the study;
8. Use of fluvoxamine, nifedipine, or warfarin for 30 days prior to Baseline Visit.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2024-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Wood, PhD, Principal Investigator — VA Puget Sound Health Care System; University of Washington
Locations (1):
- VA Puget Sound Health Care System, Tacoma, Washington, United States

REFERENCES:
- [Background] Raskind MA, Burke BL, Crites NJ, Tapp AM, Rasmussen DD. Olanzapine-induced weight gain and increased visceral adiposity is blocked by melatonin replacement therapy in rats. Neuropsychopharmacology. 2007 Feb;32(2):284-8. doi: 10.1038/sj.npp.1301093. Epub 2006 May 10. PMID 16710316

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 40 participants who were initially consented, 5 were screen fails, 13 were lost to follow up and 5 were withdrawals prior to beginning Phase I of being prescribed olanzapine. 17 participants began Phase I and 4 were lost to follow up during that phase. 13 participants went on to Phase II to be randomized to one of two melatonin groups, however 3 were not able to collect data, leaving 10 participants in Phase II.
Groups:
- Olanzapine Phase: In treatment phase I, all subjects will receive olanzapine, 10-25 mg/day.
- IIA (0.3mg/Day Melatonin): In the 0.3mg/day melatonin in treatment phase II, all subjects will receive olanzapine (10-25mg/day) plus melatonin. Subjects will be randomized at a ratio of 1:1 to receive melatonin 0.3mg/day or 3mg/day. Group IIA will receive 0.3mg/day of melatonin.
- IIB (3mg/Day Melatonin): In the 3mg/day melatonin in treatment phase II, all subjects will receive olanzapine (10-25mg/day) plus melatonin. Subjects will be randomized at a ratio of 1:1 to receive melatonin 0.3mg/day or 3mg/day. Group IIB will receive 3mg/day of melatonin.
Period: Phase I - Olanzapine Only
Arm/Group | Olanzapine Phase | IIA (0.3mg/Day Melatonin) | IIB (3mg/Day Melatonin)
Started | 17 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Period: Phase II - Randomization to Melatonin
Arm/Group | Olanzapine Phase | IIA (0.3mg/Day Melatonin) | IIB (3mg/Day Melatonin)
Started | 0 | 6 | 7
Completed | 0 | 4 | 6
Not Completed | 0 | 2 | 1
Not completed — Data unable to be collected | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IIA (0.3mg Day Melatonin) | IIB (3.0 mg/Day Melatonin) | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 6 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (6.61) | 47.33 (12.58) | 50.6 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 6 | 10
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Nocturnal Melatonin Production
Description: Nocturnal melatonin production as estimated by assay of urinary 6-sulfatoxymelatonin (aMT6s) adjusted for creatinine
Time Frame: 6 and 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IIA (0.3mg Day Melatonin) | IIB (3.0 mg/Day Melatonin)
Number analyzed (Participants) | 4 | 6
mg/dL
  Baseline | 11.19 (9.69) | 19.09 (10.12)
  Week 6 | 10.39 (8.51) | 15.18 (12.49)
  Week 12 | 197.7 (163.83) | 2,137.12 (1,430.97)

2. Secondary Outcome: Weight
Description: weight (measured in kilograms)
Time Frame: 6 weeks & 12 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | IIA (0.3mg Day Melatonin) | IIB (3.0 mg/Day Melatonin)
Number analyzed (Participants) | 4 | 6
kilograms
  Baseline | 87.10 (3.76) | 88.53 (24.99)
  Week 6 | 90.71 (3.65) | 93.20 (28.68)
  Week 12 | 93.45 (4.90) | 95.14 (28.71)

3. Secondary Outcome: Total Cholesterol
Description: Total cholesterol on metabolic blood panel
Time Frame: 6 weeks & 12 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | IIA (0.3mg Day Melatonin) | IIB (3.0 mg/Day Melatonin)
Number analyzed (Participants) | 4 | 6
mg/dL
  Baseline | 185.25 (35.68) | 204.43 (31.04)
  Week 6 | 207 (19.29) | 220.43 (29.56)
  Week 12 | 205.5 (26.01) | 221.71 (36.07)

ADVERSE EVENTS:
Groups:
- Melatonin .3mg; Melatonin 3mg: After the olanzapine phase I, participants were randomized to receive a daily dose of melatonin at either .3mg or 3 mg.
- Olanzapine Only: In phase one participants were prescribed olanzapine only
Arm/Group | Melatonin .3mg | Melatonin 3mg | Olanzapine Only
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/6 | 1/17
Other Adverse Events (participants affected / at risk) | 3/4 | 3/6 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin .3mg (N=4) | Melatonin 3mg (N=6) | Olanzapine Only (N=17)
Psychiatric Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Melatonin .3mg (N=4) | Melatonin 3mg (N=6) | Olanzapine Only (N=17)
Abnormal lab values (General disorders) | 2 (3) | 2 (2) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
Increased Blood Pressure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Psychotic symptoms (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Somnolence (General disorders) | 1 (1) | 0 (0) | 3 (3)
Tremors (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety/Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Dry mouth (General disorders) | 0 (0) | 0 (0) | 2 (2)
Flu symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1)
Increased appetite (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia/sleep disturbance (General disorders) | 0 (0) | 0 (0) | 4 (4)
Muscle pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Restless leg (General disorders) | 0 (0) | 0 (0) | 2 (2)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Results are limited by small sample size and relatively high percentage of non-completers, which diminishes the power to analyze results. Results of this small sample may not be representative of the larger population and should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No